CLINICAL TRIAL: NCT04658992
Title: A Study on the Registration of the Use of Feilike Heji in Minors
Brief Title: The Registration on the Use of Feilike Heji in Minors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhong Wang, researcher, China Academy of Chinese Medical Sciences
Other Study IDs: Feilike V2.0
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Feilike HeJi is produced by Guizhou Jianxing Pharmaceutical Co. LTD. For the treatment of phlegm heat caused by lung cough phlegm yellow, bronchial asthma, bronchitis, see the syndrome of proprietary Chinese medicine (approval number: Z20025136) approved by the state and the drug from radix scutellariae, radix peucedani, radix stemonae, red gentian root of deal, phoenix tree, spreading hedyotis herb, red tube 7 flavour, with qingrejiedu, antitussive expectorant effect. In order to fully understand the safety of Feilike HeJi in clinical practice and fulfill the responsibility of production enterprises for patients, the production enterprises initiated this study to further evaluate the safety and understanding of the function characteristics of Feilike HeJi in a wide range of people, so as to guide the clinical rational drug use.

ELIGIBILITY:
Inclusion Criteria:

* All minor patients (age <18 years old) who use Feilike Mixture at the specified monitoring time and in the monitoring center (department) .
* Voluntarily participate in this study and meet ethical requirements.

Exclusion Criteria:

* Not Applicable.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All minor patients (age <18 years old) who use Feilike Mixture at the specified monitoring time and in the monitoring center (department) and voluntarily participate in this study and meet ethical requirements.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
AE | The range of adverse events was from the beginning of the use of Feilike HeJi to 3 days after the cessation of the use of Feilike HeJi.
  All adverse events occurred during the study were determined according to CTCAE V5.0 for severity.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, Prof, Study Director — Beijing Children's Hospital affiliated to Capital Medical University
Locations (21):
- China (21):
  - Beijing Children's Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - Beijing Pinggu Hospital, Beijing, Beijing Municipality
  - Beijing Changping Hospital, Beijing, Beijing Municipality
  - Peking University Binhai Hospital, Beijing, Beijing Municipality
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Second People's Hospital of Huadu District, Guangzhou, Guangzhou, Guangdong
  - Shenzhen Pingshan Women's and Children's Health Hospital, Shenzhen, Guangdong
  - The First People's Hospital of Bijie City, Bijie, Guizhou
  - Guiyang Maternal and Child Health Hospital, Guiyang, Guizhou
  - Harbin Children's Hospital, Haerbin, Helongjiang
  - Changsha First Hospital, Changsha, Hunan
  - Xiangya San Hospital, Central South University, Changsha, Hunan
  - You County People's Hospital, Zhuzhou, Hunan
  - Second Affiliated Clinic, Nanjing Medical University, Nanjing, Jiangsu
  - Jiangxi Children's Hospital, Nanchang, Jiangxi
  - Lotus County Maternal and Child Health Hospital, Pingxiang, Jiangxi
  - Haicheng Central Hospital, Anshan, Liaoning
  - Fengcheng Central Hospital, Fengcheng, Liaoning
  - The First Hospital affiliated with The Chinese Medical University, Shenyang, Liaoning
  - Qilu Hospital, Jinan, Shandong
  - The First Affiliated Hospital of Air Force Military Medical University, Xian, Shanxi